CLINICAL TRIAL: NCT02040506
Title: A Phase 1, Open-Label Study Evaluating the Safety, Pharmacokinetics, and Clinical Activity of IGN523 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: A Phase I Study of IGN523 in Subjects With Relapsed or Refractory AML
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Igenica Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IGN523-01
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Acute Myelogenous Leukemia; Acute Myeloid Leukemia
Keywords: Acute Myelogenous Leukemia; Acute Myeloid Leukemia; Drug therapy; CD98; Relapsed; Refractory; Monoclonal antibody
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IGN523 (Experimental): IGN523
  Interventions: Drug: IGN523

INTERVENTIONS:
Drug: IGN523 — Given intravenously every week for 8 weeks. Dosing beyond 8 weeks will be permitted for subjects meeting criteria for ongoing clinical benefit and acceptable safety.

SUMMARY:
This study will examine the safety and tolerability of IGN523 administered as an IV infusion. The main purpose of the study is to determine the maximum tolerated dose (MTD), which is the highest dose that does not cause unacceptable side effects of IGN523 in patients with acute myeloid leukemia (AML). The MTD will be determined by observing the dose-limiting toxicities (the side effects that prevent further increases in dose) of IGN523. In addition, the pharmacokinetic profile and anti-leukemia activity of IGN523 will be assessed. A recommended Phase 2 dose (RP2D) of IGN523 will be identified, on the basis of safety, pharmacokinetic (PK), and pharmacodynamic (PD) data.

DETAILED DESCRIPTION:
Primary Objectives:

* Evaluate the safety and tolerability of IGN523 administered weekly
* Determine the MTD and dose limiting toxicity (DLT) of IGN523 when administered weekly during the DLT Evaluation Period
* Identify a recommended Phase 2 dose (RP2D) of IGN523 on the basis of safety, PK, and PD data

Secondary Objectives:

* Assess the incidence of antibody formation to IGN523
* Characterize the PK of IGN523 in subjects with relapsed or refractory AML
* Perform a preliminary assessment of the anti-leukemic activity of IGN523 in subjects with relapsed or refractory AML
* Perform a preliminary assessment of biologic markers that might predict IGN523 anti-leukemic activity

Estimated Enrollment: 50 Study Start Date: February 2014 Estimated Study Completion Date: March 2016 Estimated Primary Completion Date: September 2015 (Final data collection for primary outcome measure)

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or treatment-refractory AML
* Eastern Cooperative Oncology Group status 0-2
* Life expectancy of at least 12 weeks
* Adequate baseline renal and hepatic function
* Measurable disease (eg, peripheral blasts greater than 5%)

Exclusion Criteria:

* Chronic myelogenous leukemia in blast crisis
* Monoclonal therapy within 4 weeks, or chemotherapy or radiotherapy within 2 weeks
* Unresolved acute toxicity from prior anti-cancer therapy
* Prior allogeneic stem cell transplant and active graft-versus-host disease requiring systemic immunosuppressive therapy within 15 days prior to screening
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known current leptomeningeal or central nervous system (CNS) involvement of leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose

SECONDARY OUTCOMES:
Incidence of antidrug antibodies to IGN523 | Through 6 months following last dose
Blood concentrations of IGN523 | Through 6 months following last dose
Assess anti-leukemic activity of IGN523 | Initial assessment after 8 weeks of treatment
  Subjects with measurable disease will be assessed by standard criteria (Cheson). Subjects will be formally evaluated for response at the end of Cycle 2; additional evaluations may be performed during the study as clinical indicated.

CONTACTS AND LOCATIONS:
Overall Officials: William Ho, MD, PhD, Study Director — Igenica Biotherapeutics, Inc.
Locations (6):
- United States (6):
  - UCSD Medical Center / Thornton Hospital, La Jolla, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Indiana Blood and Marrow Transplantation Clinic, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - MD Anderson Cancer Center, Houston, Texas
  - University of Washington, Seattle, Washington